CLINICAL TRIAL: NCT05871359
Title: "Transcranial Direct Current Stimulation and Dual Tasks in Parkinson's Disease-tDCS&DT in PD"
Brief Title: Transcranial Direct Current Stimulation and Dual Tasks
Acronym: Tdcs&DT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Casa di Cura Privata del Policlinico SpA (Other)
Responsible Party: Principal Investigator, Paola Antoniotti, Principal Investigator, PhD candidate, Casa di Cura Privata del Policlinico SpA
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ccppdezza
Record Dates: First submitted 2023-02-06; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Transcranial direct current stimulation; Dual task; Biomarkers
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into 2 groups, using REDCap (Research Electronic Data Capture) software (Harris et al, 2009): 15 / group and will carry out activities in Dual Task (DT) associated with transcranial Direct Current Stimulation (tDCS) real (test group) or sham (control group).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tDCS group (Active Comparator): transcranial Direct Current Stimulation group (tDCS group) : patients carry out activities in Dual Task associated with tDCS real.
  Interventions: Device: Transcranial Direct Current Stimulation; Procedure: Dual task
- Sham group (Sham Comparator): Sham group: patients carry out activities in Dual Task associated with tDCS sham.
  Interventions: Device: Transcranial Direct Current Stimulation; Procedure: Dual task

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — The stimulator will be connected to two electrodes .The active electrode will be placed on the areas of the dorsal lateral pre-frontal cortex (DLPFC) contralateral to the more affected side.The other one on the supra orbital area.
Procedure: Dual task — The Dual Task consists of walking for 20 minutes along a hallway, simultaneously patient has to answer to a different ecological cognitive (attention, fluences, calculation) and motor tasks (hold a tray, turn head, ecc..)

SUMMARY:
The project aims to evaluate the clinical and biological effects on patients with Parkinson's disease of an innovative treatment characterized by the use of transcranial Direct Current Stmulation (tDCs) with Dual Task (DT), i.e. including the performance of motor activities in conjunction with the request of cognitive performance, such as executive functions (creative flexibility, working memory and divided attention).

Randomized controlled, double-blind, non-pharmacological study using device.The project involves the enrollment of 30 patients.Participants will be randomized into 2 groups: 15 / group and will carry out activities in DT associated with tDCS real (test group) or sham (control group). Each will carry out 12 rehabilitation sessions (2 / week) of 30 minutes. A follow-up is foreseen for all 12 weeks after the end of the treatment.

Patients will undergo, at baseline (T0), at the end of the session (T1) and at 12 weeks (T2), a motor and a cognitive profile, moreover a blood sample will be taken.

The project intends to improve the state of Parkinson's patients both thanks to the type of protocol that associates DT and tDCS, and thanks to the verification of the treatment through personalized biological analyzes. In detail, improvement in clinical performance, space-time variables in gait and cognitive tests are expected; the variability of synaptic and pathological markers will serve to verify the effect of the treatment.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disease characterized by motor symptoms such as tremor at rest, rigidity, bradykinesia, postural instability and cognitive deficits A growing number of studies show that transcranial direct current electrical stimulation (tDCS), a low-cost, non-invasive brain stimulation method, could potentially become a clinical tool for rehabilitation of patients with Parkinson's disease.

Furthermore, some studies have shown that walking deficit in patients with Parkinson's disease is exacerbated by adding a dual cognitive or motor task. Daily activities require walking while simultaneously performing cognitive and / or motor tasks, such as talking to a friend or carrying a glass of water. This is why there are Dual Task (DT) training programs for patients with Parkinson's disease. A recent systematic review and meta-analysis demonstrated that treatment in DT can be an effective method of improving walking in terms of walking speed and cadence, balance and other motor symptoms in patients with Parkinson's disease.

Future investigations are needed to determine stimulation characteristics and optimal dosage when combined with training in DT.

The present study aims to investigate whether the application of tDCS at the dorso lateral prefrontal cortex(DLPFC) region level can add significant improvements to the motor and cognitive profile in patients with Parkinson's disease.

Randomized controlled, double-blind, non-pharmacological study using device. The data will be collected at the Department of Neurorehabilitation Sciences of the Polyclinic Nursing Home in Milan.

The project involves the enrollment of 30 patients. Each patient will take part in the study after an overall assessment of the general medical conditions, in relation to the suitability for participation in the study, by the neurologist of the unit department of Neuromotor Rehabilitation.

Randomized quadruple-blind study in parallel groups, in which the therapist who will carry out the treatment and the patient will not be aware of the assignment to the group (experimental vs control). Participants will be randomized into 2 groups, using Research Electronic Data Capture (RedCap) software:15 / group and will carry out activities in DT associated with tDCS real (test group) or sham (control group). Each will carry out 12 rehabilitation sessions (2 / week) of 30 minutes. A follow-up is foreseen for all 12 weeks after the end of the treatment.

Patients will undergo, at baseline (T0), at the end of the session (T1) and at 12 weeks (T2), a motor and a cognitive profile, moreover a blood sample will be taken.

The project intends to improve the state of Parkinson's patients both thanks to the type of protocol that associates DT and tDCS, and thanks to the verification of the treatment through personalized biological analyzes. In detail, improvement in clinical performance, space-time variables in gait and cognitive tests are expected; the variability of synaptic and pathological markers will serve to verify the effect of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease patient (Hoehn and Yahr I-III);
* Ability to walk with or without aid for 100 meters,
* Mini Mental State Examination> 21,
* Ability to express informed consent

Exclusion Criteria:

* Inability of the patient to understand or perform the task based on the evaluation and judgment of the referring neuropsychologist and the investigator, and / or to sign or initial the informed consent;
* History of other previous, disabling neurological diseases (e.g., Stroke cerebri, Alzheimer's Disease, Multiple Sclerosis and Disabling Peripheral Neuropathy) and / or ongoing psychiatric diseases (e.g., major depression);
* Presence of contraindications to stimulation according to the most recent guidelines;
* Brain metal implants- Pace-makers, brain stimulators, cochlear implants- Pregnancy status (for women);
* Patient denial of informed consent.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2025-09-12 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Change of duration (seconds) of 10 Meters Walking Test (single and dual task) | At baseline (t0) after 45 days (t1) and after 84 days (t2)
  Patient has to walk for ten meters with (dual task) or without(single task) a cognitive task
Change of duration (seconds) of Time Up and Go (single and dual task) | At baseline (t0) after 45 days (t1) and 84 days (t2)
  Patient has to sit from a chair, walk for 3 meters, turn and walk back to sit on the chair, with (dual task) or without (single task) a cognitive task.

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS; part III-motor part) | At baseline, after 45 days (t1) and 84 days (t2)
  Assessment on motor performance (balance, walking, manual dexterity) UPDRS, the minimum value is 0,the maximum is 132, higher scores mean worse outcome.
Mini-best test, | At baseline (t0),after 45 days (t1) and 84 days (t2)
  Assessment of balance, the minimum value is 0,the maximum is 28, higher scores mean better outcome.
Freezing Of Gait questionnaire (FOG) | At baseline (t0),after 45 days (t1) and 84 days (t2)
  Assessment of freezing of gait .The minimum value is 0,the maximum is 24, higher scores mean worse outcome.
Montreal Cognitive Assessment (MoCA; Conti et al., 2015) | At baseline (t0), after 45 days (t1) and 84 days (t2)
  Index of global cognitive and executive functioning
Digit Span Forward e Backward (Monaco et al. 2013) | At baseline (t0),after 45 days (t1) and 84 days (t2)
  The assessment of short-term and verbal working memory
Wisconsin Card Sorting Test (Laiacona et al., 2000) | At baseline (t0),after 45 days (t1) and 84 days (t2)
  To assess planning, flexibility and monitoring skills in a complex problem-solving task
Trail Making Test (TMT; Giovagnoli et al., 1996) | At baseline (t0),after 45 days (t1) and 84 days (t2)
  Processing speed index and attentional shifting
Italian version of the Parkinson's Disease-Cognitive Rating Scale (PD-CRS; Santangelo et al., 2014). | At baseline (t0),after 45 days (t1) and 84 days (t2)
  Tests for the assessment of immediate verbal memory, visual comparison naming, sustained attention, working memory, clock drawing, deferred verbal memory, alternating fluency, verbal fluency of actions
Biomarkers (Brain Derived Neurotrophic Factor BDNF, dopamine, synaptic proteins, α-synuclein, inflammatory and oxidative stress factors, circRNA, miRNA, with techniques of biochemistry, genetics and immunohistochemistry) | At baseline (t0),after 45 days (t1) and 84 days (t2)
  A blood sample will be taken to acquire plasma, serum and exosomes.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Corbo, Study Director — Department of Neurological Science Casa di Cura del Policlinico
Locations (1):
- Dipartimento di scienze neuroriabilitative, Casa di Cura del Policlinico, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antal A, Alekseichuk I, Bikson M, Brockmöller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Flöel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9): Appollonio I, Leone M, Isella V et al (2005) The frontal assessment battery (FAB): normative values in an Italian population sample. Neurol Sci 26:108-116. Barbarotto, R., Laiacona, M., Frosio, R. et al. A normative study on visual reaction times and two Stroop colour-word tests. Ital J Neuro Sci 19, 161-170 (1998). Beck, A.T., Steer, R.A., & Brown, G.K. (1996). Manual for the Beck Depression Inventory-II. San Antonio, TX: Psychological Corporation. Bloem BR, Marinus J, Almeida Q, Dibble L, Nieuwboer A, Post B, Ruzicka E, Goetz C, Stebbins G, Martinez-Martin P, Schrag A, Movement Disorders Society Rating Scales C Measurement instruments to assess posture, gait, and balance in Parkinson's disease: Critique and recommendations. Mov Disord. 2016. Broeder S, Nackaerts E, Heremans E, Vervoort G, Meesen R, Verheyden G, et al. Transcranial direct current stimulation in Parkinson's disease: neurophysiological mechanisms and behavioral effects. Neurosci Biobehav Rev. 2015. Caffarra, P., Vezzadini, G., Dieci, F., Zonato, F., & Venneri, A. (2002). Una versione abbreviata del test di Stroop: Dati normativi nella popolazione Italiana. Nuova Rivista di Neurologia, 12(4), 111-115. Carlesimo, G. A., Buccione, I., Fadda, L., Graceffa, A., Mauri, M., Lorusso, S., Bevilacqua, G., & Caltagirone, C. (2002). Standardizzazione di due test di memoria per uso clinico: Breve Racconto e Figura di Rey. Nuova Rivista di Neurologia, 12(1), 1-13. Costa A, Bagoj E, Monaco M, Zabberoni S, De Rosa S, Papantonio AM, Mundi C, Caltagirone C, Carlesimo GA. Standardization and normative data obtained in the Italian population for a new verbal fluency instrument, the phonemic/semantic alternate fluency test. Neurol Sci. 2014 Mar;35(3):365-72. doi: 10.1007/s10072-013-1520-8. Epub 2013 Aug 21. PMID: 23963806. Conti S, Bonazzi S, Laiacona M, Masina M, Coralli MV. Montreal Cognitive Assessment (MoCA)-Italian version: regression based norms and equivalent scores. Neurol Sci. 2015 Feb;36(2):209-14. doi: 10.1007/s10072-014-1921-3. Epub 2014 Aug 20. PMID: 25139107. Christopher G. Goetz,1 * Barbara C. Tilley,2 Stephanie R. Shaftman,2 Glenn T. Stebbins,1 Stanley Fahn,3 Pablo Martinez-Martin,4 Werner Poewe,5 Cristina Sampaio,6 Matthew B. Stern,7 Richard Dodel,8 Bruno Dubois,9 Robert Holloway,10 Joseph Jankovic,11 Jaime Kulisevsky,12 Anthony E. Lang,13 Andrew Lees,14 Sue Leurgans,1 Peter A. LeWitt,15 David Nyenhuis,16 C. Warren Olanow,17,18 Olivier Rascol,19 Anette Schrag,20 Jeanne A. Teresi,21 Jacobus J. van Hilten,22 and Nancy LaPelle,23 for the Movement Disorder Society UPDRS Revision Task Forc. Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Scale Presentation and Clinimetric Testing Results. MOVEMENT DISORDER,2008. Cho SS, Strafella AP. rTMS of the left dorsolateral prefrontal cortex modulates dopamine release in the ipsilateral anterior cingulate cortex and orbitofrontal cortex. PLoS One. 2009 Aug 21;4(8):e6725. doi: 10.1371/journal.pone.0006725. PMID: 19696930; PMCID: PMC2725302. Fregni F, Boggio PS, Santos MC, Lima M, Vieira AL, Rigonatti SP, et al. Noninvasive cortical stimulation with transcranial direct current stimulation in Parkinson's disease. Mov Disord. 2006;21(10):1693-702. Felipe Fregni, MD, PhD, Mirret M. El-Hagrassy, MD, Kevin Pacheco-Barrios, MD, MSc, Sandra Carvalho, PhD, Jorge Leite, PhD, Marcel Simis, MD, PhD, Jerome Brunelin, PhD, Ester Miyuki Nakamura-Palacios, MD, PhD, Paola Marangolo, PhD, Ganesan Venkatasubramanian, MD, PhD, Daniel San-Juan, MD, PhD, Wolnei Caumo, MD, PhD, Marom Bikson, PhD, André R. Brunoni, MD, PhD, and Neuromodulation Center Working Group. Evidence-based guidelines and secondary meta-analysis for the use of transcranial direct current stimulation (tDCS) in neurological and psychiatric disorders, 2021.